CLINICAL TRIAL: NCT04383470
Title: Collaborative Outcomes Study on Health and Functioning During Infection Times During COVID-19 Pandemic
Acronym: COH-FIT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Padova (Other)
Collaborators: Northwell Health (Other); Donald and Barbara Zucker School of Medicine at Hofstra/Northwell (Unknown)
Responsible Party: Sponsor
Other Study IDs: COH-FIT
Record Dates: First submitted 2020-04-27; First posted 2020-05-12 (Actual); Last update posted 2020-05-14 (Actual); Status verified 2020-05

CONDITIONS: Mental Health Wellness 1; Pandemic
Keywords: COVID-19; Mental Health; Physical Health; Infection; Resilience
MeSH Terms: conditions — COVID-19; Psychological Well-Being; Infections

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- General population, during COVID pandemic: General population during COVID-19 pandemic. Adults, adolescents, and children aged 6 years or older. People working in health-care, police, fire-, and military-service vs others. People with physical illness vs others. People with mental illness vs others. Different continents, countries, and regions.
- General population, 6 months after COVID pandemic: General population, 6 months after COVID pandemic Adults, adolescents, and children aged 6 years or older. People working in health-care, police, fire-, and military-service vs others. People with physical illness vs others. People with mental illness vs others. Different continents, countries, and regions.
- General population, 12 months after COVID pandemic: General population, 12 months after COVID pandemic Adults, adolescents, and children aged 6 years or older. People working in health-care, police, fire-, and military-service vs others. People with physical illness vs others. People with mental illness vs others. Different continents, countries, and regions.

SUMMARY:
Observational, cross-sectional, multi-center, multi-wave survey, assessing characteristics and predictors of physical and mental health as well as health behaviors during COVID-19 pandemic, targeting the general population (children, adolescents and adults).

DETAILED DESCRIPTION:
In March 2020, the World Health Organization declared the COVID-19 (known as Coronavirus) virus a global pandemic. COVID-19 is a variant of coronavirus thought to originate in Wuhan province China. Up until April 7, 2020, as many as 1,346,299 individuals had confirmed COVID-19 infection, with already 74,679 deaths from COVID-19 complications.

The hypothesis of this study is that the physical and mental health of the general population and health care workers involved in the management of COVID-19 infected people is heavily affected by COVID-19, but that risk and protective factors exist.

Investigators plan to distribute 3 different surveys based on the age group. The first survey, COH-FIT-Adults/ (COH-FIT-A), will be distributed the general adult (age >/= 18 years old) population in North America, South America, Europe, Asia, Africa and Australia via an online link, making the general population aware of the project via public announcements, social media and regular media coverage outlets, or via specialized institutes and agencies (e.g., opinion research centers) that are capable of using a randomly selected, nationally representative sample (potentially funded by national / local grant applications). For the subgroup of adult health-care professionals, additionally, survey distribution mechanisms will be used that utilize medical professional organizations and associations, hospital and university anonymized channels.

Guardians of adolescents aged 14-17 years old will be asked to provide electronic consent for their adolescent to participate in the COH-FIT-AD survey after having taken the survey and being familiar with the questions, being informed that the one question having sexuality as the content will be omitted from the adolescent version. Guardians of children aged 6-13 years old will be able to review the survey questions that children would answer before electronically consenting to participate.

ELIGIBILITY:
Inclusion Criteria:

* General population
* Consenting to the study (adults)
* Guardians consenting to study participation of children and adolescents

Exclusion Criteria:

* Not consenting to the study (adults)
* Not assenting to the study (children and adolescents)
* age < 6 years old

Min Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: General population
Sampling Method: Non-Probability Sample
Enrollment: 100000 (Estimated)
Dates: Start 2020-04-26 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Mental health symptoms, well-being change from last 2 weeks before the pandemic to last 2 weeks during COVID-19 pandemic | wave 1 - change from last 2 weeks before pandemic to the following from April 26th 2020 on, until the pandemic will be over as declared by WHO (we estimate between October 2020 and April 2021)
  Primary outcome in the wave 1 survey, conducted during the COVID-19 pandemic, will be mean change in visual analogue scale-assessed transdiagnostic measures across all psychiatric symptoms, and World Health Organization (WHO)-5 well-being in the last 2 weeks compared to the last 2 weeks of "regular life" before the COVID-19 outbreak.
  For WHO-5 the raw score ranges from 0 (absence of well-being) to 25 (maximal well-being).
Mental health symptoms, well-being change from last 2 weeks before the pandemic to last 2 weeks 6 months after WHO declares pandemic over COVID-19 pandemic | wave 2 - change from before to 6 months after pandemic
  Primary outcome in the wave 2 survey, conducted during the COVID-19 pandemic, will be mean change in visual analogue scale-assessed transdiagnostic measures across all psychiatric symptoms and World Health Organization (WHO)-5 well-being in the last 2 weeks six months after the COVID-19 pandemic ended, compared to the last 2 weeks of "regular life" before the COVID-19 outbreak.
  For WHO-5 the raw score ranges from 0 (absence of well-being) to 25 (maximal well-being).
Mental health symptoms change, well-being change from last 2 weeks before the pandemic to last 2 weeks 12 months after WHO declares pandemic over COVID-19 pandemic | wave 3 - change from before to 12 months after pandemic (after the pandemic outbreak has been declared from WHO, and until the pandemic outbreak has been declared conlucded by WHO)
  Primary outcome in the wave 3 survey, conducted during the COVID-19 pandemic, will be mean change in visual analogue scale-assessed transdiagnostic measures across all psychiatric symptoms and World Health Organization (WHO)-5 well-being in the last 2 weeks 12 months after the COVID-19 pandemic ended, compared to the last 2 weeks of "regular life" before the COVID-19 outbreak.
  For WHO-5 the raw score ranges from 0 (absence of well-being) to 25 (maximal well-being).

SECONDARY OUTCOMES:
Change in alcohol abuse, as change in units used from last 2 weeks before the pandemic to last 2 weeks during pandemic | wave 1 - change from last 2 weeks before pandemic to the following from April 26th 2020 on, until the pandemic will be over as declared by WHO (we estimate between October 2020 and April 2021)
  Change in alcohol abuse, as change in units used from last 2 weeks before the pandemic to last 2 weeks during pandemic
Change in cigarettes use, as change in number of cigarettes per day from last 2 weeks before the pandemic to last 2 weeks during pandemic | wave 1 - change from last 2 weeks before pandemic to the following from April 26th 2020 on, until the pandemic will be over as declared by WHO (we estimate between October 2020 and April 2021)
  Change in cigarettes use, as change in number of cigarettes per day from last 2 weeks before the pandemic to last 2 weeks during pandemic
Change in grams of cannabinoids smoked from last 2 weeks before the pandemic to last 2 weeks during pandemic | wave 1 - change from last 2 weeks before pandemic to the following from April 26th 2020 on, until the pandemic will be over as declared by WHO (we estimate between October 2020 and April 2021)
  Change in grams of cannabinoids smoked from last 2 weeks before the pandemic to last 2 weeks during pandemic
Change in alcohol abuse, as change in units used from last 2 weeks before the pandemic to last 2 weeks during pandemic | wave 2 - change from before to 6 months after pandemic
  Change in alcohol abuse, as change in units used from last 2 weeks before the pandemic to last 2 weeks during pandemic
Change in cigarettes use, as change in number of cigarettes per day from last 2 weeks before the pandemic to last 2 weeks during pandemic | wave 2 - change from before to 6 months after pandemic
  Change in cigarettes use, as change in number of cigarettes per day from last 2 weeks before the pandemic to last 2 weeks during pandemic
Change in grams of cannabinoids smoked from last 2 weeks before the pandemic to last 2 weeks during pandemic | wave 2 - change from before to 6 months after pandemic
  Change in grams of cannabinoids smoked from last 2 weeks before the pandemic to last 2 weeks during pandemic
Change in alcohol abuse, as change in units used from last 2 weeks before the pandemic to last 2 weeks during pandemic | wave 3 - change from before to 12 months after pandemic
  Change in alcohol abuse, as change in units used from last 2 weeks before the pandemic to last 2 weeks during pandemic
Change in cigarettes use, as change in number of cigarettes per day from last 2 weeks before the pandemic to last 2 weeks during pandemic | wave 3 - change from before to 12 months after pandemic
  Change in cigarettes use, as change in number of cigarettes per day from last 2 weeks before the pandemic to last 2 weeks during pandemic
Change in grams of cannabinoids smoked from last 2 weeks before the pandemic to last 2 weeks during pandemic | wave 3 - change from before to 12 months after pandemic
  Change in grams of cannabinoids smoked from last 2 weeks before the pandemic to last 2 weeks during pandemic
Change in general physical health, self-rated, on a VAS scale from 0 to 100. | wave 1 - change from last 2 weeks before pandemic to the following from April 26th 2020 on, until the pandemic will be over as declared by WHO (we estimate between October 2020 and April 2021)
  Change in general physical health, self-rated, on a VAS scale from 0 to 100.
Change in general physical health, self-rated, on a VAS scale from 0 to 100. | wave 2 - change from before to 6 months after pandemic
  Change in general physical health, self-rated, on a VAS scale from 0 to 100.
Change in general physical health, self-rated, on a VAS scale from 0 to 100. | wave 3 - change from before to 12 months after pandemic
  Change in general physical health, self-rated, on a VAS scale from 0 to 100.
Change in general mental health, self-rated, on a VAS scale from 0 to 100. | wave 1 - change from last 2 weeks before pandemic to the following from April 26th 2020 on, until the pandemic will be over as declared by WHO (we estimate between October 2020 and April 2021)
  Change in general mental health, self-rated, on a VAS scale from 0 to 100.
Change in general mental health, self-rated, on a VAS scale from 0 to 100. | wave 2 - change from before to 6 months after pandemic
  Change in general mental health, self-rated, on a VAS scale from 0 to 100.
Change in general mental health, self-rated, on a VAS scale from 0 to 100. | wave 3 - change from before to 12 months after pandemic
  Change in general mental health, self-rated, on a VAS scale from 0 to 100.
Change in easiness of access to care, self-rated a on a VAS scale from 0 to 100. | wave 1 - change from last 2 weeks before pandemic to the following from April 26th 2020 on, until the pandemic will be over as declared by WHO (we estimate between October 2020 and April 2021)
  Change in easiness of access to care, self-rated a on a VAS scale from 0 to 100.
Change in easiness of access to care, self-rated a on a VAS scale from 0 to 100. | wave 2 - change from before to 6 months after pandemic
  Change in easiness of access to care, self-rated a on a VAS scale from 0 to 100.
Change in easiness of access to care, self-rated a on a VAS scale from 0 to 100. | wave 3 - change from before to 12 months after pandemic
  Change in easiness of access to care, self-rated a on a VAS scale from 0 to 100.
Change in medication adherence, self-rated a on a VAS scale from 0 to 100. | wave 1 - change from last 2 weeks before pandemic to the following from April 26th 2020 on, until the pandemic will be over as declared by WHO (we estimate between October 2020 and April 2021)
  Change in medication adherence, self-rated a on a VAS scale from 0 to 100.
Change in medication adherence, self-rated a on a VAS scale from 0 to 100. | wave 2 - change from before to 6 months after pandemic
  Change in medication adherence, self-rated a on a VAS scale from 0 to 100.
Change in medication adherence, self-rated a on a VAS scale from 0 to 100. | wave 3 - change from before to 12 months after pandemic
  Change in medication adherence, self-rated a on a VAS scale from 0 to 100.
Change in functioning in self-care, school/work, social, and family, self-rated a on a VAS scale from 0 to 100. | wave 1 - change from last 2 weeks before pandemic to the following from April 26th 2020 on, until the pandemic will be over as declared by WHO (we estimate between October 2020 and April 2021)
  Change in functioning in self-care, school/work, social, and family, self-rated a on a VAS scale from 0 to 100.
Change in functioning in self-care, school/work, social, and family, self-rated a on a VAS scale from 0 to 100. | wave 2 - change from before to 6 months after pandemic
  Change in functioning in self-care, school/work, social, and family, self-rated a on a VAS scale from 0 to 100.
Change in functioning in self-care, school/work, social, and family, self-rated a on a VAS scale from 0 to 100. | wave 3 - change from before to 12 months after pandemic
  Change in functioning in self-care, school/work, social, and family, self-rated a on a VAS scale from 0 to 100.

CONTACTS AND LOCATIONS:
Overall Officials: Christoph U. Correll, MD, Principal Investigator — Northwell Health; Marco Solmi, MD, Principal Investigator — University of Padova; Agorastos Agorastos, MD, Study Director — Aristotle University Of Thessaloniki; Andres Estradè, MSc, Study Director — Universidad Católica del Uruguay
Locations (1):
- Aristotle University of Thessaloniki, Thessaloniki, Greece

REFERENCES:
- [Derived] Agorastos A, Thompson T, Solmi M, Cortese S, Estrade A, Radua J, Dragioti E, Vancampfort D, Thygesen LC, Aschauer H, Schlogelhofer M, Aschauer E, Schneeberger A, Huber CG, Hasler G, Conus P, Do Cuenod KQ, von Kanel R, Arrondo G, Fusar-Poli P, Gorwood P, Llorca PM, Krebs MO, Scanferla E, Kishimoto T, Rabbani G, Skonieczna-Zydecka K, Brambilla P, Favaro A, Takamiya A, Zoccante L, Colizzi M, Bourgin J, Kaminski K, Moghadasin M, Seedat S, Matthews E, Wells J, Vassilopoulou E, Gadelha A, Su KP, Kwon JS, Kim M, Lee T, Papsuev O, Mankova D, Boscutti A, Gerunda C, Saccon D, Righi E, Monaco F, Croatto G, Cereda G, Demurtas J, Brondino N, Veronese N, Enrico P, Politi P, Ciappolino V, Pfennig A, Bechdolf A, Meyer-Lindenberg A, Kahl KG, Domschke K, Bauer M, Koutsouleris N, Winter SM, Borgwardt S, Bitter I, Balazs J, Czobor P, Unoka Z, Mavridis D, Tsamakis K, Bozikas VP, Tunvirachaisakul C, Maes M, Rungnirundorn T, Supasitthumrong T, Haque A, Brunoni AR, Costardi CG, Schuch FB, Polanczyk G, Luiz JM, Fonseca L, Aparicio LV, Valvassori SS, Nordentoft M, Vendsborg P, Hoffmann SH, Sehli J, Sartorius N, Heuss SC, Guinart D, Hamilton J, Kane J, Rubio J, Sand M, Koyanagi A, Solanes A, Andreu-Bernabeu A, Caceres ASJ, Arango C, Diaz-Caneja CM, Hidalgo-Mazzei D, Vieta E, Gonzalez-Penas J, Fortea L, Parellada M, Fullana MA, Verdolini N, Andrlikova E, Janku K, Millan MJ, Honciuc M, Moniuszko-Malinowska A, Loniewski I, Samochowiec J, Kiszkiel L, Marlicz M, Sowa P, Marlicz W, Spies G, Stubbs B, Firth J, Sullivan S, Darcin AE, Aksu H, Dilbaz N, Noyan O, Kitazawa M, Kurokawa S, Tazawa Y, Anselmi A, Cracco C, Machado AI, Estrade N, De Leo D, Curtis J, Berk M, Carvalho AF, Ward P, Teasdale S, Rosenbaum S, Marx W, Horodnic AV, Oprea L, Alexinschi O, Ifteni P, Turliuc S, Ciuhodaru T, Bolos A, Matei V, Nieman DH, Sommer I, van Os J, van Amelsvoort T, Sun CF, Guu TW, Jiao C, Zhang J, Fan J, Zou L, Yu X, Chi X, de Timary P, van Winkel R, Ng B, Pena E, Arellano R, Roman R, Sanchez T, Movina L, Morgado P, Brissos S, Aizberg O, Mosina A, Krinitski D, Mugisha J, Sadeghi-Bahmani D, Sheybani F, Sadeghi M, Hadi S, Brand S, Errazuriz A, Crossley N, Ristic DI, Lopez-Jaramillo C, Efthymiou D, Kuttichira P, Kallivayalil RA, Javed A, Afridi MI, James B, Seb-Akahomen OJ, Fiedorowicz J, Daskalakis J, Yatham LN, Yang L, Okasha T, Dahdouh A, Tiihonen J, Shin JI, Lee J, Mhalla A, Gaha L, Brahim T, Altynbekov K, Negay N, Nurmagambetova S, Jamei YA, Weiser M, Correll CU. Mental health, coping and related risk factors during the first 2 years of the COVID-19 pandemic in children: Nationally representative, multi-wave, cross-sectional results from 12 countries from the global COH-FIT study. Eur Neuropsychopharmacol. 2025 Dec 18;104:112741. doi: 10.1016/j.euroneuro.2025.112741. Online ahead of print. PMID 41418519
- See also: COH-FIT Survey — https://neuroscienze.unipd.it/redcap/surveys/?s=WW7CH8HEHJ